CLINICAL TRIAL: NCT06494969
Title: Effect of Sevoflurane Versus Total Intravenous Anesthesia on Intraocular Pressure in Patients Undergoing Coronary Artery Bypass Graft Surgery With Cardiopulmonary Bypass: A Prospective Observational Study
Brief Title: Intraocular Pressure in Patients Undergoing Coronary Artery Bypass Graft Surgery With Cardiopulmonary Bypass
Status: Completed | Type: Observational
Sponsor: Antalya Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: Yasemin1
Record Dates: First submitted 2024-06-28; First posted 2024-07-10 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-05

CONDITIONS: Intraocular Pressure; Anesthesia
Keywords: Intraocular pressure; cardiac surgery; coronary artery bypass grafting
MeSH Terms: interventions — Tonometry, Ocular

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group P: Propofol-based total intravenous anesthesia
  Interventions: Device: Intraocular pressure measurement
- Group S: Sevoflurane-based anesthesia
  Interventions: Device: Intraocular pressure measurement

INTERVENTIONS:
Device: Intraocular pressure measurement — Intraocular pressures were measured and recorded at 8 predefined time points using a tonometer; before anesthesia induction (T1), 10 min after induction (T2), immediately before the beginning of CPB (T3), 3 minute after the beginning of CPB (T4), 3 minute after cross-clamping (T5), 3min after cross-clamp removal (T6), immediately before the weaning of CPB (T7), and end of the surgery (immediately after skin closure) (T8).

SUMMARY:
The aim of the study to compare the effects of sevoflurane-based anesthesia and propofol-based total intravenous anesthesia on intraocular pressure (IOP) during coronary artery bypass graft surgery (CABG) with cardiopulmonary bypass (CPB).

The primary endpoint was to examine the effects of propofol-based total intravenous anesthesia (TIVA) and sevoflurane-based anesthesia methods on IOP during CABG operation. Secondary endpoints included a comparison of hemodynamic variables, blood gas values, intensive care, and hospital stay.

DETAILED DESCRIPTION:
Patients undergoing elective coronary artery bypass grafting surgery with cardiopulmonary bypass (CPB) were included in this prospective observational study. Patients with a history of cardiac surgery, diabetic retinopathy, cataract, uncontrolled hypertension, chronic kidney disease, glaucoma, previous eye surgery, previous neurological disease, allergy to propofol or sevoflurane, and a baseline intraocular pressure (IOP) greater than 30 mmHg were excluded from the study. The primary endpoint was to examine the effects of propofol-based total intravenous anesthesia (TIVA) and sevoflurane-based anesthesia methods on IOP during CABG operation. Secondary endpoints included a comparison of hemodynamic variables, blood gas values, intensive care, and hospital stay.

Intraoperative anesthesia management was standardized for both techniques, and the attending anesthesiologist was asked to comply with the protocols determined within the scope of this standardization. However, the choice between sevoflurane-based anesthesia or propofol-based TIVA was left to the discretion of the attending cardiac anesthesiologists. In the operating theatre, patients were monitored with a 5-lead electrocardiography, invasive arterial blood pressure via radial artery catheterization, pulse oximetry, and rectal temperature. Initial vital signs and blood gas values were recorded. No premedication was given before anesthesia induction. Anesthesia induction was performed in all patients with intravenous administration of 0.1 mg/kg midazolam, 5-10 mcg/kg fentanyl, 0.5-2 mg/kg propofol, and 0.6 mg/kg rocuronium. An endotracheal tube with an internal diameter of 8-8.5 mm was used for male patients and an endotracheal tube with an internal diameter of 7-7.75 mm for female patients. Mechanical ventilation was performed using a Drager Perseus anesthesia workstation under volume-controlled mode, with fractional inspired oxygen tension (Fio2) set at 0.5, positive end-expiratory pressure (PEEP) at 4-5 cmH2O, tidal volume at 6-8 ml/kg of predicted body weight, and respiratory rate adjusted to maintain end-tidal carbon dioxide (EtCO2) between 35-45 mmHg. A central venous catheter was inserted into all patients using the right internal jugular vein after induction, and a Foley catheter was inserted for urine monitoring. Depth of anesthesia was monitored in all patients using Patient State Index (PSI) values (Masimo®, Masimo Corporation, Irvine, CA, USA), and PSI values were maintained between 25-50 throughout the surgery in all patients. Rocuronium was administered as 0.1-0.2 mg/kg IV intermittent bolus doses for muscle relaxation.

According to the choice of anesthesia type, the patients were divided into two groups: those using propofol-based total intravenous anesthesia (TIVA) (Group P) and those using sevoflurane-based anesthesia (Group S). In Group P, anesthesia was maintained with an infusion of 3-10 mg/kg/h IV propofol. In Group S, anesthesia maintenance was provided with 1-1.5 minimum alveolar concentration (MAC) sevoflurane. In both groups, fentanyl was administered if the increase in mean arterial pressure (MAP) was greater than 20% from the baseline but not less than 65 mmHg. During CPB in Group S, sevoflurane was delivered to the oxygenator circuit via a calibrated vaporizer (Blease®, Blease Medical Equipment, Ltd, Chesham, UK), and the MAC value was measured at the oxygenator output of the CPB circuit. Extracorporeal circulation was provided with a CPB device (Stockert®, Sorin Group, Munchen, Germany) and an oxygenator (Sechrist®, Sechrist Int, Anaheim, CA, USA). Before CPB, 300-400 U/kg heparin was administered to achieve an Activated Coagulation Time (ACT) of 480 s. During CPB, non-pulsatile flow with a target flow rate of 2.2-2.5 l/min/m2 was applied, and body temperature was maintained between 32-34°C. Hematocrit values were maintained between at least 20-25%, and mean arterial pressure at 50-80 mmHg. Myocardial protection was maintained with intermittent antegrade and sometimes retrograde blood cardioplegia. Before weaning from CPB, patients were warmed to 36-37°C, and heparin was neutralized with 1 mg IV protamine sulfate per 100 U. All patients were transferred to the cardiovascular surgery intensive care unit (ICU) without extubation after the operation.

Intraocular pressures were measured at eight predefined time points using the ICARE Tonometer (Icare Finland Oy, Vantaa, Finland) by a single ophthalmologist blinded to group allocation (Table 1). Three consecutive measurements were taken from each eye at each time point, and the average value of IOP for each eye was recorded.

Arterial blood gas values (pH, PO2, PCO2, lactate, and hematocrit) were recorded at three different time points: Before induction, during CPB (after cross-clamping), and at the end of the surgery. In addition, hemodynamic variables (systolic, diastolic, and mean arterial pressures, heart rate, and SpO2 values) were recorded at the same time points as IOP measurements. The length of hospital stay and ICU stay of the patients were also recorded.

I n conclusion intraocular pressures were similar for both groups at all time points. A statistically significant decrease was found in intraocular pressures in all measurements after induction compared to pre-induction values in both Group P and Group S (p < 0.05). Compared to IOP measured at 10 minutes after induction, no statistically significant difference was found at all subsequent time points in both groups. When the right and left intraocular pressures were compared, no statistically significant difference was detected at all time points in both Group P and Group S.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective coronary artery bypass grafting surgery with cardiopulmonary bypass (CPB)

Exclusion Criteria:

* history of cardiac surgery
* diabetic retinopathy
* cataract
* uncontrolled hypertension
* chronic kidney disease
* glaucoma
* previous eye surgery
* previous neurological disease
* allergy to propofol or sevoflurane
* baseline intraocular pressure (IOP) greater than 30 mmHg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective coronary artery bypass grafting surgery with cardiopulmonary bypass (CPB) were included.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-01-03 (Actual); Study Completion 2022-01-28 (Actual)

PRIMARY OUTCOMES:
Intraocular pressure during coronary artery bypass graft surgery with cardiopulmonary bypass | Through study completion, an average of 6 months
  Examine the effects of propofol based total intravenous anesthesia and sevoflurane-based anesthesia methods on intraocular pressure during coronary artery bypass graft surgery operation

CONTACTS AND LOCATIONS:
Overall Officials: Ali Sait Kavaklı, Study Director — Associate professor
Locations (1):
- Health Science University, Antalya Training and Research Hospital, Antalya, Muratpasa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No